CLINICAL TRIAL: NCT04590911
Title: Effectiveness of Multimodal Cognitive Rehabilitation for Traumatic Brain Injury Sustained During Older Adulthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Michelle McKerral, Professor and Researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRIR
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: TBI (Traumatic Brain Injury); Rehabilitation; Aging
Keywords: traumatic brain injury; cognitive rehabilitation; aging; memory; executive functions; psychological well-being; daily life activities
MeSH Terms: conditions — Brain Injuries, Traumatic; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Semi-randomized, controlled, before-after study with follow-up at six-months with blinded outcome measurement
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEP intervention (Experimental): Cognitive Enrichment Program (CEP) : tailored for individuals who sustain a TBI in later adulthood. The CEP is a 12-week multimodal intervention structured into three modules designed to simultaneously address cognitive problems resulting from TBI, as well as age-related cognitive issues in the following domains: self-awareness, attention and memory, and executive functions.
  Interventions: Behavioral: Cognitive Enrichment Program (CEP)
- Usual care (No Intervention): Usual care : interventions within a holistic interdisciplinary rehabilitation program focused on resuming daily activities and social roles, if needed, as determined by treating physician; does not include any form of cognitive rehabilitation.

INTERVENTIONS:
Behavioral: Cognitive Enrichment Program (CEP) — Multimodal cognitive rehabilitation program for individuals having sustained a traumatic brain injury during older adulthood
  Arms: CEP intervention

SUMMARY:
In a worldwide context of accelerated demographic aging, traumatic brain injury (TBI) in older adults has become a public health problem. TBI incidence grows following an exponential curve as people get older, increasing the occurrence of TBI in ageing individuals. Rehabilitation programs used in clinical settings have generally been developed for younger adults, and their efficacy with older adults who sustain a TBI has not been evaluated. The investigators have tailored a modular cognitive rehabilitation program for individuals who sustain a TBI in older adulthood, the Cognitive Enrichment Program (CEP), by adapting approaches which have shown to be effective in normal ageing and with other neurological conditions. The aim of the study is to evaluate the effectiveness of the CEP in adults having sustained a TBI during later adulthood. Specific objectives are to evaluate the effectiveness on memory, executive functions, psychological well-being and daily life activities using psychometric tests, self-reported questionnaires, and daily life-like tasks. The investigators hypothesize that memory and executive functions training included in the CEP will result in an improvement in both psychometric and self-reported scores in a trained group of older individuals with TBI, whereas this will not be the case for a comparable TBI group who did not receive the CEP intervention.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of a multimodal cognitive intervention, the Cognitive Enrichment Program (CEP), on episodic memory, executive functions, psychological well-being and daily life activities in traumatic brain injured (TBI) older adults, as compared to an active control group that receives only usual care in the form of holistic rehabilitation. The experimental design is a semi-randomized, controlled, before-after study with blinded outcome measurement. French-speaking participants aged 55 years or older and having sustained a mild, moderate or severe TBI at least 6 months before enrollment, were recruited by clinical coordinators from one hospital and from two outpatient interdisciplinary rehabilitation centres. The CEP consists of three intervention modules, Introduction and self-awareness, Attention and Memory, and Executive functions, which were conducted with groups of 5 participants, in 90-minute sessions, twice weekly, during 12 weeks. The CEP was conducted by an experienced clinical neuropsychologist. Assessments of intervention effects were performed by trained evaluators, who were blinded to group assignment of participants, in two separate sessions lasting about 90 minutes each. There were three assessment time-points: baseline (pre-intervention - T0); 14-weeks (post-intervention - T1); 6-months post-intervention (follow-up - T2). Primary outcome measures (neuropsychological and self-report) were chosen to measure targeted effects of the CEP and generalization measures (self-report) were used to evaluate broader effects of the intervention. Control measures were also used to control for spontaneous recovery.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with mild, moderate or severe TBI at least six months before enrolment in study, based on the World Health Organization criteria [16]: Mild: length of loss or altered level of consciousness (LOC) 0-30 minutes, Glasgow Coma Scale (GCS) score 13-15/15, negative or positive brain imaging (CT-Scan or MRI), post-traumatic amnesia (PTA) duration <24 hrs; Moderate: LOC 30 min-24 hrs, GCS score 9-12, positive brain imaging, PTA duration 1-14 days; Severe: LOC >24 h, GCS score 3-8, positive brain imaging, PTA duration >2 weeks [16];
2. post-traumatic amnesia period must be already resolved;
3. aged at least 55 years;
4. fluent in French (speaking, understanding, reading).

Exclusion Criteria:

1. previously received or receiving another specific or direct cognitive intervention focusing on similar or identical cognitive functions;
2. diagnosis or documented clinical impressions of dementia (medical files) or Montreal Cognitive Assessment score lower than 20;
3. diagnosis of an active psychiatric condition;
4. consumption of alcohol (drinking 5 or more drinks on the same occasion on each of 5 or more days weekly in the past 30 days), or consuming illicit drugs.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline (T0) Face-name association (Côte-des-Neiges Computerized Memory Battery) at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Episodic memory measure where participants have to associate 12 previously learned face-name pairs.
Change from post-intervention (T1) Face-name association (Côte-des-Neiges Computerized Memory Battery) at 6 months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Episodic memory measure where participants have to associate 12 previously learned face-name pairs.
Change from baseline (T0) Word list recall (Côte-des-Neiges Computerized Memory Battery) at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Episodic memory measure where participants have to associate 12 previously learned words. Measures of immediate and delayed recall were obtained.
Change from post-intervention (T1) Word list recall (Côte-des-Neiges Computerized Memory Battery) at 6-months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Episodic memory measure where participants have to associate 12 previously learned words. Measures of immediate and delayed recall were obtained.
Change from baseline (T0) Text memory (Côte-des-Neiges Computerized Memory Battery) at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Episodic memory measure where participants have to recall a short text, which is divided into 23 macrostructure elements (main ideas of the text giving a meaning to the story), and 24 microstructure elements (specific details about the story). Measures of immediate and delayed recall were obtained for macrostructure and microstructure elements.
Change from post-intervention (T1) Text memory (Côte-des-Neiges Computerized Memory Battery) at 6-months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Episodic memory measure where participants have to recall a short text, which is divided into 23 macrostructure elements (main ideas of the text giving a meaning to the story), and 24 microstructure elements (specific details about the story). Measures of immediate and delayed recall were obtained for macrostructure and microstructure elements.
Change from baseline (T0) Self-Evaluation Memory Questionnaire (SEMQ) at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Self-report memory measure where participants rate (1 to 6; never to always) their memory performance for 10 dimensions for which are derived mean scores: Conversations, Books & movies, Slips of attention, People, Use of objects, Political & social events, Places, Actions to perform, Personal events, General. Higher scores indicate worse outcome.
Change from post-intervention (T1) Self-Evaluation Memory Questionnaire (SEMQ) at 6-months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Self-report memory measure where participants rate (1 to 6; never to always) their memory performance for 10 dimensions for which are derived mean scores: Conversations, Books & movies, Slips of attention, People, Use of objects, Political & social events, Places, Actions to perform, Personal events, General. Higher scores indicate worse outcome.
Change from baseline (T0) Six Elements Task-Adapted (SET-A) at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Executive function measure where participants complete a task where the goal is to earn as many points as possible while following specific rules. Five dimensions are rated according to the degree of attainment (0-3) : Tackling the 6 subtasks, Inter-task balance, Avoiding rule-breaking, Checking time at appropriate moments, and Efficient behavior. The Total score (/15) is also computed.
Change from post-intervention (T1) Six Elements Task-Adapted (SET-A) at 6-months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Executive function measure where participants complete a task where the goal is to earn as many points as possible while following specific rules. Five dimensions are rated according to the degree of attainment (0-3) : Tackling the 6 subtasks, Inter-task balance, Avoiding rule-breaking, Checking time at appropriate moments, and Efficient behavior. The Total score (/15) is also computed.
Change from baseline (T0) Sorting Test - Delis-Kaplan Executive Function System (D-KEFS) at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Executive function measure where participant must sort cards with printed words into groups in as many ways as possible and describe their sorting criteria. Measures used are: Confirmed Correct Sort Total (CCS) raw score, Free Sorting Description (FSD) total raw score, and Time-Per-Sort Ratio (TSR) in seconds.
Change from post-intervention (T1) Sorting Test - Delis-Kaplan Executive Function System (D-KEFS) at 6-months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Executive function measure where participant must sort cards with printed words into groups in as many ways as possible and describe their sorting criteria. Measures used are: Confirmed Correct Sort Total (CCS) raw score, Free Sorting Description (FSD) total raw score, and Time-Per-Sort Ratio (TSR) in seconds.
Change from baseline (T0) Stroop Test - Four-color version at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Executive function measure where participant complete four tasks (reading, colors, inhibition and flexibility). The measures used (time, in seconds) are Inhibition of the Stroop effect by verbally indicating the color of the ink instead of reading the words, and Flexibility, where participants indicate the color of the ink and read the words when they appear in a box.
Change from post-intervention (T1) Stroop Test - Four-color version at 6-months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Executive function measure where participant complete four tasks (reading, colors, inhibition and flexibility). The measures used (time, in seconds) are Inhibition of the Stroop effect by verbally indicating the color of the ink instead of reading the words, and Flexibility, where participants indicate the color of the ink and read the words when they appear in a box.
Change from baseline (T0) Dysexecutive Questionnaire (DEX) at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Self-report executive function measure where participants rate (0 to 5; never to always) their executive functioning on three scales: Executive cognition, Behavioural-Emotional Self-Regulation, and Metacognition. Self-awareness of executive difficulties was used as a measure of generalization by calculating the difference between participants' and a significant other's scores on the three subscales. Higher scores indicate worse outcome.
Change from post-intervention (T1) Dysexecutive Questionnaire (DEX) at 6-months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Self-report executive function measure where participants rate (0 to 5; never to always) their executive functioning on three scales: Executive cognition, Behavioural-Emotional Self-Regulation, and Metacognition. Self-awareness of executive difficulties was used as a measure of generalization by calculating the difference between participants' and a significant other's scores on the three subscales. Higher scores indicate worse outcome.
Change from baseline (T0) Psychological General Well-Being Index (PGWBI) at 14 weeks (post-intervention - T1) | 14 weeks (pre-post intervention - T0-T1)
  Self-report measure where participants rate (0-6; low to high) their self-perceived well-being on 22 items. Higher scores indicate better outcome.
Change from post-intervention (T1) Psychological General Well-Being Index (PGWBI) at 6-months post-intervention (follow-up - T2) | 6-months post-intervention (follow-up - T2)
  Self-report measure where participants rate (0-6; low to high) their self-perceived well-being on 22 items. Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McKerral, PhD, Principal Investigator — CRIR-IURDPM-CCSMTL and Université de Montréal
Locations (1):
- Iurdpm-Ccsmtl, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cisneros E, de Guise E, Belleville S, McKerral M. A controlled clinical efficacy trial of multimodal cognitive rehabilitation on episodic memory functioning in older adults with traumatic brain injury. Ann Phys Rehabil Med. 2021 Sep;64(5):101563. doi: 10.1016/j.rehab.2021.101563. Epub 2021 Aug 5. PMID 34325040
- [Derived] Cisneros E, Beausejour V, de Guise E, Belleville S, McKerral M. The impact of multimodal cognitive rehabilitation on executive functions in older adults with traumatic brain injury. Ann Phys Rehabil Med. 2021 Sep;64(5):101559. doi: 10.1016/j.rehab.2021.101559. Epub 2021 Aug 5. PMID 34303000